CLINICAL TRIAL: NCT01866514
Title: A Study Evaluating Use of the Proximal Humerus Intraosseous Vascular Access Site for Anesthesia Patient Positioning
Brief Title: Proximal Humerus Site for Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013-07
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2013-05

CONDITIONS: Intraosseous Vascular Access
Keywords: EZ-IO; IO; Intraosseous Vascular Access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anesthesia Arm (Experimental): proximal humerus intraosseous vascular access will be established bilaterally in the proximal humerus using the anesthesia approach in which the arm is abducted from the body.
  Interventions: Procedure: proximal humerus intraosseous vascular access; Drug: 2% preservative-free lidocaine; Device: EZ-IO

INTERVENTIONS:
Procedure: proximal humerus intraosseous vascular access — The arm receiving the IO needle is positioned with the arm abducted to shoulder level (in position required for surgery), with the arm rotated inward, into the optimal position, with the palms faced down. Deeply palpate the humerus until the junction of the humeral shaft and the humeral head, the surgical neck is identified; the insertion site is in the surgical neck. With the 45mm IO needle placed perpendicular to the plane of the skin, the IO needle is inserted into the surgical neck using a slightly superior angle of insertion and the needle is inserted to the hub. The stylet will be removed and an EZ-Connect primed with 2% preservative-free lidocaine will be attached to the catheter hub. Aspirate return will be attempted to confirm needle placement within the medullary cavity.
  Other Names: EZ-IO; Instraosseous Access; Proximal Humerus intraosseous access; IO access; proximal humerus IO access
Drug: 2% preservative-free lidocaine
Device: EZ-IO

SUMMARY:
This will be a prospective, non-controlled study using healthy adult volunteers as subjects receiving bilateral proximal humerus intraosseous (IO) vascular access to evaluate the insertion technique and IO infusion flow rates.

DETAILED DESCRIPTION:
When using IO access in the perioperative and OR settings, abduction of the arms to the shoulder level prevents use of the traditional proximal humerus insertion site due to the rotation of the humeral head under the acromion process. An alternate proximal humerus IO insertion technique has been developed to meet the needs of anesthesia patient positioning that uses a slightly more distal insertion site and a superior angle of insertion. However infusion flow rate in the proximal humerus using the anesthesia technique has not been measured. This study is needed to evaluate the anesthesia proximal humerus IO insertion technique to determine if the IO infusion flow rates remain unchanged by the alternate method.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older Have no amputation of the upper extremities Able to lay flat on table for up to 2 hours Self-reported as healthy, as confirmed by the PI

Exclusion Criteria:

* Have an active infection in the body Imprisoned Pregnant Cognitively impaired Fracture in humerus, or significant trauma to the site Excessive tissue and/or absence of adequate anatomical landmarks in humerus Infection in target area Humeral IO insertion in past 48 hours, prosthetic limb or joint or other significant orthopedic procedure in humerus Current use of anti-coagulants Current cardiac condition requiring pacemaker or anti-arrhythmic drugs Prior adverse reaction to lidocaine

Volunteers with any of the following characteristics may be excluded from the infusion pathway evaluation involving administration of contrast dye at the discretion of the PI.

Prior adverse reaction to contrast dye Allergy to any food or drug History of impaired renal function History of impaired hepatic function History of cardiac disease History of pheochromocytoma

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Intraosseous Infusion Flow rate | Day 1 after establishing proximal humerus IO vascular access
  The primary objective of the study is to evaluate the infusion flow rates attainable when using the anesthesia approach to establish proximal humerus IO vascular access.
  The primary endpoints will be the infusion flow rate obtained at each tested infusion pressure, including gravity, 100 mmHg, 200 mmHg, and 300 mmHg.

SECONDARY OUTCOMES:
Evaluate relationship between IO and peripheral venous blood | Day 1 after establishing proximal humerus IO vascular access and peripheral venous access
  The secondary objectives for this study are to evaluate the relationship between IO and peripheral venous blood when used for routine laboratory testing.
  Secondary Endpoints will include results of routine blood analysis.
The secondary objective for this study is to evaluate the infusion pathway from the proximal humerus to the heart. | Day 1 after establishing proximal humerus intraosseous vascular access
  The secondary objectives for this study is to evaluate the infusion pathway from the proximal humerus.
  Secondary Endpoint will be time in seconds for fluid delivery from the proximal humerus to the heart, using visualization of contrast injection under fluoroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Larry J Miller, MD, Principal Investigator — Vidacare Corporation
Locations (1):
- Bulverde-Spring Branch EMS, Spring Branch, Texas, United States